CLINICAL TRIAL: NCT05949138
Title: Clinical Data Collection and Evaluation of ECG-Less Cardiac CT
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Collaborators: University of Chicago (Other); University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: 11771729874
Record Dates: First submitted 2023-06-14; First posted 2023-07-17 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Cardiac CT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- ECG-Less Cardiac CT: Enrolled subjects will receive a clinically-indicated, diagnostic Cardiac CT with contrast. No ECG leads will be applied.
  Interventions: Device: ECG-Less Cardiac CT using SmartPhase

INTERVENTIONS:
Device: ECG-Less Cardiac CT using SmartPhase — Administration of medications and biologic products (such as contrast agent administration, and potentially beta-blockers and other medications) will be given according to standard hospital care.
  This is a prospective research study evaluating an investigational workflow on an existing CT device that has regulatory clearance. The investigational workflow includes preforming the CT acquisition according to the hospital's usual care with the exception that the ECG signal which triggers the scan will be coming from an ECG simulator based on an estimate of the patient's heart rate, rather than through ECG leads connected to the subject. Clinically-indicated Cardiac CTs take approximately 30-60 minutes. No additional imaging is needed as part of the study.

SUMMARY:
The primary objective of this study is to collect CT scan data without ECG-leads attached to the human subject. This data is intended to represent a typical range of clinical scenarios in which Cardiac CT imaging is used.

DETAILED DESCRIPTION:
Data collected in this study will be used for technology development, scientific evaluation, marketing and education, and regulatory submissions for future products. This is a pre-market, prospective, open-label, non-randomized, single arm data collection clinical study conducted at one site in the United States of America.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be included in this study if they meet the following criteria:

1. Who are 18 year of age or older;
2. Able to sign and date the informed consent form; AND
3. Who are scheduled for a clinical-indicated Cardiac CT exam that will include contrast administration.

Exclusion Criteria:

Subjects may be excluded from participating in study if they meet any of the following criteria:

1. Who are pregnant or lactating;
2. Who were previously enrolled in this study;
3. Anyone with known or suspected allergy to iodinated contrast agents;
4. Anyone with known or suspected renal insufficiency as determined by site medical personnel;
5. Who are scheduled for a CT cardiac calcium scoring test;
6. Who are in need of urgent or emergent care;
7. Who have any conditions that, in the opinion of the PI or designee, would interfere with the evaluation of the results or constitute a health hazard for the subject; AND
8. Who are unwilling to have GEHC personnel present for the CT exam.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population will consist of adults that are 18-years of age or older, and who are scheduled for a clinically indicated cardiac CT exam that will include contrast administration.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Data Collection | Through study completion, an average of 6 months
  Number of Participants with raw investigational cardiac CT scan data

CONTACTS AND LOCATIONS:
Overall Officials: Kayla Matcheck, Study Director — GE Healthcare
Locations (2):
- United States (2):
  - University of Chicago, Chicago, Illinois
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No